CLINICAL TRIAL: NCT02274558
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel, Fixed-Dose Study to Assess the Efficacy, Safety, and Tolerability of NBI-98854 for the Treatment of Tardive Dyskinesia
Brief Title: A Phase 3 Study of NBI-98854 for the Treatment of Tardive Dyskinesia
Acronym: KINECT 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-1304
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NBI-98854 40 mg (Experimental): NBI-98854 administered as one (1) 40 mg capsule and one (1) placebo capsule, taken by mouth, every morning between 7:00am - 10:00am for 6 weeks. At the end of Week 6, subjects will enter a double-blind NBI-98854 treatment period and continue with their current dose.
  Interventions: Drug: NBI-98854; Drug: Placebo
- NBI-98854 80 mg (Experimental): Subjects randomized to the NBI-98854 80 mg dose will receive NBI-98854 40 mg for the first week (administered as one (1) 40 mg capsule and one (1) placebo capsule), followed by NBI-98854 80 mg administered as two (2) 40 mg capsules, taken by mouth, every morning between 7:00am - 10:00am for 5 weeks. At the end of Week 6, subjects will enter a double-blind NBI-98854 treatment period and continue with their current dose.
  Interventions: Drug: NBI-98854; Drug: Placebo
- Placebo (Experimental): Placebo administered as two (2) placebo capsules, taken by mouth, every morning between 7:00am - 10:00am for 6 weeks. At the end of Week 6, subjects will enter a double-blind NBI-98854 treatment period and be randomized to either a 40 mg or 80 mg dose. Subjects re-randomized to receive NBI-98854 80 mg will receive 40 mg for the first week.
  Interventions: Drug: NBI-98854; Drug: Placebo

INTERVENTIONS:
Drug: NBI-98854 — NBI-98854 40 mg capsules
Drug: Placebo — NBI-98854 placebo capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of NBI-98854 administered once daily for the treatment of Tardive Dyskinesia (TD) symptoms.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel, fixed-dose study to evaluate the efficacy, safety, and tolerability of two doses of NBI-98854 (40 mg and 80 mg) compared to placebo, administered once daily. The study design includes a double-blind, placebo-controlled treatment period for 6 weeks and a double-blind NBI-98854 treatment period for an additional 42 weeks, for a total of 48 weeks of treatment. Final follow-up assessments will be conducted 4 weeks after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study.
2. Female subjects must not be pregnant.
3. Have one of the following clinical diagnoses for at least 3 months prior to screening: Schizophrenia or Schizoaffective Disorder, or Mood Disorder.
4. Have a clinical diagnosis of neuroleptic-induced TD for at least 3 months prior to screening.
5. Have moderate or severe TD.
6. If using maintenance medication(s) for schizophrenia or schizoaffective disorder, or mood disorder, be on stable doses.
7. Be in good general health.
8. Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.
9. Have a negative drug screen for amphetamines,barbiturates, benzodiazepines, phencyclidine, cocaine, opiates, or cannabinoids

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening.
2. Have a known history of substance dependence, or substance (drug) or alcohol abuse
3. Have a significant risk of suicidal or violent behavior.
4. Have a known history of neuroleptic malignant syndrome.
5. Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
6. Have a cancer diagnosis within 3 years of screening (some exceptions allowed)
7. Have received an investigational drug within 30 days prior to screening or plan to use an investigational drug (other than NBI-98854) during the study.
8. Have a blood loss ≥550 mL or donated blood within 30 days prior to Baseline.
9. Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
10. Have had previous exposure with NBI-98854 or had previously participated in an NBI-98854 clinical study.
11. Are currently pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Principal Investigator — Neurocrine Biosciences
Locations (54):
- United States (48):
  - Little Rock, Arkansas
  - Anaheim, California
  - Glendale, California
  - Irvine, California
  - Long Beach, California
  - Los Angeles, California
  - National City, California
  - Norwalk, California
  - Oakland, California
  - Oceanside, California
  - San Bernardino, California
  - San Diego, California
  - Torrance, California
  - Bradenton, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Leesburg, Florida
  - Maitland, Florida
  - Miami, Florida
  - North Miami, Florida
  - Chicago, Illinois
  - Oak Brook, Illinois
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Amherst, New York
  - Cedarhurst, New York
  - Rochester, New York
  - Durham, North Carolina
  - Pinehurst, North Carolina
  - Dayton, Ohio
  - Shaker Heights, Ohio
  - Oklahoma City, Oklahoma
  - Conshohocken, Pennsylvania
  - Norristown, Pennsylvania
  - Phoenixville, Pennsylvania
  - Scranton, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - DeSoto, Texas
  - Fort Worth, Texas
  - Irving, Texas
  - Petersburg, Virginia
  - Spokane, Washington
- Canada (4):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Puerto Rico (2):
  - Caguas
  - San Juan

REFERENCES:
- [Derived] Sajatovic M, Alexopoulos GS, Burke J, Farahmand K, Siegert S. The effects of valbenazine on tardive dyskinesia in older and younger patients. Int J Geriatr Psychiatry. 2020 Jan;35(1):69-79. doi: 10.1002/gps.5218. Epub 2019 Oct 31. PMID 31617235
- [Derived] Correll CU, Cutler AJ, Kane JM, McEvoy JP, Liang GS, O'Brien CF. Characterizing Treatment Effects of Valbenazine for Tardive Dyskinesia: Additional Results From the KINECT 3 Study. J Clin Psychiatry. 2018 Dec 18;80(1):18m12278. doi: 10.4088/JCP.18m12278. PMID 30695293
- [Derived] Factor SA, Remington G, Comella CL, Correll CU, Burke J, Jimenez R, Liang GS, O'Brien CF. The Effects of Valbenazine in Participants with Tardive Dyskinesia: Results of the 1-Year KINECT 3 Extension Study. J Clin Psychiatry. 2017 Nov/Dec;78(9):1344-1350. doi: 10.4088/JCP.17m11777. PMID 29141124
- [Derived] Grigoriadis DE, Smith E, Hoare SRJ, Madan A, Bozigian H. Pharmacologic Characterization of Valbenazine (NBI-98854) and Its Metabolites. J Pharmacol Exp Ther. 2017 Jun;361(3):454-461. doi: 10.1124/jpet.116.239160. Epub 2017 Apr 12. PMID 28404690
- [Derived] Hauser RA, Factor SA, Marder SR, Knesevich MA, Ramirez PM, Jimenez R, Burke J, Liang GS, O'Brien CF. KINECT 3: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial of Valbenazine for Tardive Dyskinesia. Am J Psychiatry. 2017 May 1;174(5):476-484. doi: 10.1176/appi.ajp.2017.16091037. Epub 2017 Mar 21. PMID 28320223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with schizophrenia or schizoaffective disorder with tardive dyskinesia (TD) or mood disorder with TD from 63 centers in North America and Puerto Rico. The last patient completed in August 2016.
Groups:
- Placebo-Controlled Placebo: Participants received Placebo capsule (matching valbenazine capsules) once daily for 6 weeks.
- Placebo-Controlled Valbenazine 40mg: Participants received valbenazine 40mg capsule once daily for 6 weeks.
- Placebo-Controlled Valbenazine 80mg: Participants received valbenazine 40mg capsule once daily for 1 week, then 80mg capsule once daily for 5 weeks.
Period: Overall Study
Arm/Group | Placebo-Controlled Placebo | Placebo-Controlled Valbenazine 40mg | Placebo-Controlled Valbenazine 80mg
Started | 78 | 76 | 80
Included in the Safety Analysis Set | 76 | 72 | 79
Completed | 71 | 63 | 71
Not Completed | 7 | 13 | 9
Not completed — Adverse Event | 2 | 4 | 2
Not completed — Non-compliance | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 4
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Included all subjects who were randomized to a treatment group and dispensed study drug, with the following 2 exclusions: (a) subjects who withdrew from the study and returned all previously dispensed study drug with all doses present, and (b) subjects who had no postbaseline safety data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Controlled Placebo | Placebo-Controlled Valbenazine 40mg | Placebo-Controlled Valbenazine 80mg | Total
Number analyzed (Participants) | 76 | 72 | 79 | 227
Age, Continuous [Mean (Full Range); unit: years] | 57.0 [30 to 84] | 55.3 [26 to 74] | 56.0 [32 to 83] | 56.1 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 40 | 104
  Male | 42 | 42 | 39 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  American Indian or Alaska Native, Caucasian | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 0 | 1
  Black or African American | 29 | 26 | 32 | 87
  Caucasian | 43 | 41 | 44 | 128
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other: Arabic | 1 | 0 | 0 | 1
  Other: Hispanic | 0 | 0 | 1 | 1
  Other: Mexican | 1 | 1 | 0 | 2
  Other: Mixed | 1 | 1 | 0 | 2
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.03 [18.1 to 42.2] | 28.64 [19.4 to 40.6] | 27.78 [18.2 to 46.9] | 28.13 [18.1 to 46.9]
Psychiatric Diagnosis Category [Count of Participants; unit: Participants]
  Schizophrenia/Schizoaffective disorder | 50 | 48 | 52 | 150
  Mood disorder | 26 | 24 | 27 | 77
Age at TD Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some subjects.
  years
    number analyzed (Participants) | 54 | 50 | 58 | 162
    (all) | 49.4 [29 to 81] | 47.8 [22 to 67] | 47.6 [17 to 72] | 48.2 [17 to 81]
BPRS Total Score [Mean (Full Range); unit: units on a scale] — The Brief Psychiatric Rating Scale (BPRS) is a clinician-rated tool designed to assess change in the severity of psychopathology in patients with schizophrenia and other psychotic disorders (Overall and Gorham, 1962, 1988). The severity of each of the 18 items of the BPRS is rated on a scale of 1 (not present) to 7 (extremely severe) (total score range: 18 to 126). Higher scores represent greater symptom severity.
  units on a scale | 29.3 [18 to 46] | 30.6 [20 to 48] | 29.1 [18 to 48] | 29.7 [18 to 48]
Baseline AIMS Total Dyskinesia Score [Mean (Standard Deviation); unit: units on a scale] — The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
  units on a scale | 9.9 (4.3) | 9.7 (4.1) | 10.4 (3.6) | 10.0 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score Change From Baseline at Week 6
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by blinded central AIMS video raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline and Week 6
Population: Intent to treat (ITT) analysis set (all subjects in the safety analysis set who have a baseline (Day -1) AIMS dyskinesia total score value and at least one post-randomization AIMS dyskinesia total score value reported during the placebo-controlled treatment period).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo: Participants received Placebo capsule (matching valbenazine capsules) once daily for 6 weeks.
- Valbenazine 80mg: Participants received valbenazine 40mg capsule once daily for 1 week, then 80mg capsule once daily for 5 weeks.
- Valbenazine 40mg: Participants received valbenazine 40mg capsule once daily for 6 weeks.
Arm/Group | Placebo | Valbenazine 80mg | Valbenazine 40mg
Number analyzed (Participants) | 69 | 70 | 63
scores on a scale | -0.1 (0.4) | -3.2 (0.4) | -1.9 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 80mg; Control for multiplicity was accomplished through the a fixed-sequence testing procedure for Week 6 outcomes: * AIMS dyskinesia total score mean change from baseline (CFB): valbenazine 80 mg vs. placebo. * CGI-TD mean score: VBZ 80 mg vs. PBO. * AIMS: VBZ 40 mg vs. PBO. * CGI-TD: VBZ 40 mg vs. PBO. For a test result in the above list to be considered statistically significant, all of the test results higher in the list must have been significant at the 0.05 level of significance; Test type: Other; p < 0.0001, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-4.2 to -2.0], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 40mg; Test type: Other; p = 0.0021, Mixed-effect Model Repeated Measures — Nominal P-value, not adjusted for multiplicity. See comments in above statistical analysis overview regarding the fixed-sequence testing procedure to control for multiplicity; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.0 to -0.7], Standard Error of Mean 0.6

2. Secondary Outcome: Clinical Global Impression of Change - TD (CGI-TD) at Week 6
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Valbenazine 40mg | Valbenazine 80mg
Number analyzed (Participants) | 69 | 63 | 70
scores on a scale | 3.2 (0.1) | 2.9 (0.1) | 2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 40mg; Test type: Other; p = 0.0742, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 80mg; Test type: Other; p = 0.0560, Mixed-effect Model Repeated Measures; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.0], Standard Error of Mean 0.1

3. Secondary Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score Responder Analysis at Week 6
Description: Percentage of AIMS responders (subjects who had at least a 50 percent reduction in AIMS score from baseline)
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Valbenazine 40mg | Valbenazine 80mg
Number analyzed (Participants) | 69 | 63 | 70
Participants | 6 | 15 | 28
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 40mg; Test type: Other; p = 0.0200, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 80mg; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Placebo | Valbenazine 40mg | Valbenazine 80mg
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/72 | 1/79
Serious Adverse Events (participants affected / at risk) | 3/76 | 4/72 | 6/79
Other Adverse Events (participants affected / at risk) | 7/76 | 9/72 | 5/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Valbenazine 40mg (N=72) | Valbenazine 80mg (N=79)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hostility (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Valbenazine 40mg (N=72) | Valbenazine 80mg (N=79)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.